CLINICAL TRIAL: NCT02931786
Title: Does Magnetic Resonance Imaging Increase Core Body Temperature in Anesthetized Children? Evaluating the Effects of Propofol and Ketofol
Brief Title: Effects of Propofol and Ketofol on Core Body Temperature in MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr Cigdem Akyol Beyoğlu, medical specialist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 118099
Record Dates: First submitted 2016-02-19; First posted 2016-10-13 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2017-11

CONDITIONS: Children
Keywords: core body temperature; magnetic resonance imaging; propofol; ketofol
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol (Active Comparator): body core temperature was measured from tympanic membrane after 1 mg/kg propofol administration, before and after magnetic resonance imaging
  Interventions: Drug: propofol; Drug: Ketamine propofol mixture
- ketofol (Active Comparator): body core temperature was measured from tympanic membrane after 0,1 ml/kg administration of ketamine propofol mixture of 10 mg/ml both, before and after magnetic resonance imaging
  Interventions: Drug: propofol; Drug: Ketamine propofol mixture

INTERVENTIONS:
Drug: propofol — propofol, midazolam and atropine administration via intravenous cannula.
  Other Names: propofol 1%
Drug: Ketamine propofol mixture — Administration of ketamine propofol mixture, midazolam and atropine via intravenous cannula
  Other Names: ketofol

SUMMARY:
Investigators researched the effect of two different types of drugs on core body temperature during magnetic resonance imaging. The hypothesis is in ketamine group, thermo disregulation is not as distinct as in propofol group, due to its positive effect on thermo regulation

DETAILED DESCRIPTION:
Intravenous anesthetics may impair thermoregulation. Absorption of radiofrequency waves by the body surface may result in heating, especially in small children during magnetic resonance imaging (MRI). Investigators applied two different intravenous anesthetics as propofol and ketamine and studied the effect of these drugs on core body temperature.

All patients aged between 6 months-10 years were administered midazolam and atropine. After that 1 mg/ kg of propofol was applied in group I, and 0,1 ml/kg of propofol ketamine mixture ( 10 mg/ml each) was applied in group II. Core body temperatures were taken before and after MRI and compared.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 6 months-10 years,
* underwent MRI under anesthesia
* ASA I-II

Exclusion Criteria:

* History of drug allergy
* Severe pulmonary and cardiac disease
* Intracranial hypertension

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in core body temperature | during magnetic resonance imaging (MRI) procedure
  temperature was taken from tympanic membrane bilaterally before and after MRI. If temperature change was more or les than 0.1 degrees celsius the patient was considered as warmer or cooler.

IPD SHARING:
Plan to Share IPD: No